CLINICAL TRIAL: NCT01343225
Title: Pilot Study of the Effect of a Non-tenofovir, Non-efavirenz-based HIV Regimen on Bone Density and Vitamin D Levels in African-American Patients With HIV Infection
Brief Title: Effect of a Non-tenofovir, Non-efavirenz-based HIV Regimen on Bone Density and Vitamin D Levels in African-American Patients With HIV Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: East Carolina University (Other)
Responsible Party: Paul Cook, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IISP # 38879
Record Dates: First submitted 2011-04-26; First posted 2011-04-28 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: HIV
Keywords: African american vitamin d bone density; African American male or female treatment naive
MeSH Terms: interventions — Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- atripla (Active Comparator): comparator
  Interventions: Drug: atripla
- darunavir ritonavir raltegravir (Experimental): experimental
  Interventions: Drug: darunavir ritonavir raltegravir

INTERVENTIONS:
Drug: atripla — once a day
  Arms: atripla
Drug: darunavir ritonavir raltegravir — as directed
  Arms: darunavir ritonavir raltegravir

SUMMARY:
2. Objectives

1. To determine the vitamin D status of African-American HIV patients who are HIV-treatment naïve.
2. To compare the effects of an efavirenz-containing regimen to a protease inhibitor regimen on 25-hydroxyvitamin D and 1,25 dihydroxyvitamin D3 levels.
3. To compare the effect on bone density of a tenofovir- and efavirenz-containing regimen to a regimen that does not contain these drugs.
4. To compare the efficacy of an alternative regimen (raltegravir, darunavir, ritonavir) to a standard once-daily regimen (tenofovir-emtricitabine-efavirenz).

Hypothesis

The investigators hypothesize that patients receiving efavirenz will be more likely to have lower 25-hydroxyvitamin D and 1,25 dihydroxyvitamin D3levels based on the fact that efavirenz is an inducer of CYP3A4 and CYP24 enzymes that degrade 25-hydroxyvitamin D and 1,25 dihydroxyvitamin D3, respectively, to inactive metabolites. The investigators speculate that patients on a tenofovir-containing regimen will be more likely to have progression of bone density loss compared to those in the non-tenofovir-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 50 years old
* HIV infection and HIV RNA > 4000 copies/ml of plasma

Exclusion Criteria:

* known risks for osteoporosis, including low body mass index (BMI < 20)
* chronic alcohol use
* chronic steroid use
* use of phenytoin or phenobarbital
* chronic renal insufficiency (calculated glomerular filtration rate < 50 ml/min)
* males with testosterone deficiency, and post-menopausal females will be excluded

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Vitamin D levels and bone density | 48 weeks
  collection of vitamin d levels and bone density measured before and at end of 48 weeks

SECONDARY OUTCOMES:
viral load and CD 4 count | 48 weeks
  Viral load and CD 4 at baseline and 48 weeks